CLINICAL TRIAL: NCT01330485
Title: Deficits in Emotion Regulation Skills as a Maintaining Factor in Major Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Friedrich-Alexander-Universität Erlangen-Nürnberg (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Matthias Berking, Ph.D., Prof. Dr., Friedrich-Alexander-Universität Erlangen-Nürnberg
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: BE4510/3-1
Record Dates: First submitted 2011-04-04; First posted 2011-04-07 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Major Depressive Disorder
Keywords: depression; emotion regulation; affect regulation; skills; randomized controlled trial; mediation
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Emotional Regulation; Negotiating

STUDY DESIGN:
Intervention Model Description: Group (3 groups) x time
Who Masked: Outcomes Assessor
Masking Description: Assessors were blinded to study conditions.
Oversight: Data Monitoring Committee: No

ARMS (3):
- Affect Regulation Training (Experimental): Affect Regulation Training as described in Berking & Whitley, 2014.
  Interventions: Behavioral: Affect Regulation Training
- Common Factor Control Condition (CFC) (Active Comparator): Common factor based therapy control condition
  Interventions: Behavioral: Common Factor Control Condition
- Waitlist Control Condition (No Intervention): Wait List Control

INTERVENTIONS:
Behavioral: Affect Regulation Training — The ART is a transdiagnostic, group-based intervention that has been developed to explicitly target emotion regulation skills (e.g., the abilities to be aware of, understand, accept, tolerate and modify negative emotions).
  Other Names: ART
  Arms: Affect Regulation Training
Behavioral: Common Factor Control Condition — The CFC is an active treatment condition designed to control for unspecific effects of psychotherapeutic interventions.
  Other Names: CFC
  Arms: Common Factor Control Condition (CFC)

SUMMARY:
The primary aim of the study is to evaluate the efficacy of a systematic training of general affect regulation skills (ART) on the reduction of depressive symptom in individuals meeting criteria for major depressive disorder (MDD).

DETAILED DESCRIPTION:
Deficits in general emotion regulation skills have been shown to be associated with various mental disorders. Thus, general affect-regulation training has been proposed as promising transdiagnostic approach to the treatment of psychopathology. In the present study, we aimed to evaluate the efficacy of a general affect-regulation as a stand-alone, group-based treatment for depression. For this purpose, we randomly assigned 218 individuals who met criteria for major depressive disorder (MDD) to the Affect Regulation Training (ART), to a waitlist control condition (WLC), or to a condition controlling for common factors (CFC). The primary outcome was the course of depressive symptom severity as assessed with the Hamilton Rating Scale for Depression and the Beck Depression Inventory. Differences between groups will be analyzed with the help of multi-level analyses. To clarify mechanisms of change we will test whether changes in emotion regulation skills will mediate potential differences between conditions regarding change of depressive symptoms. As secondary goal, the study will try and clarify whether participating in ART might augment the efficacy of subsequent individual cognitive-behavioral therapy.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of MDD according to DSM-IV criteria as the primary diagnosis
* age 18 and above
* sufficient German language skills

Exclusion Criteria:

* high risk of suicide
* indication of substantial secondary gain
* currently in psychotherapeutic treatment with an institution/professional other than those involved in the study
* co-occurring psychotic, bi-polar, and/or substance disorders
* organic brain disorder(s), severe medical condition, and/or severe cognitive impairment that impedes ability to participate in the study or treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2010-11; Primary Completion 2014-04 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change in depressive symptoms | Pre to post ART, CFC or WLC; hence covering the ten week time period from the first assessment point (prior to randomization) to the assessment point 10 weeks later
  Change in depressive symptoms as assessed in Beck Depression Inventory (BDI-II) and Hamilton Rating Scale for Depression (HRSD) and aggregated to a composite score is possible

SECONDARY OUTCOMES:
Emotion regulation skills | Pre to post ART, CFC or WLC; hence covering the ten week time period from the first assessment point (prior to randomization) to the assessment point 10 weeks later
  Emotion regulation skills as assessed with the Emotion Regulation Skills Questionnaire

OTHER OUTCOMES:
General psychopathological symptom load | Pre to post ART, CFC or WLC; hence covering the ten week time period from the first assessment point (prior to randomization) to the assessment point 10 weeks later
  General psychopathological symptom load as assessed with the Brief Symptom Inventory
Course of depressive symptoms during individual CBT after ART/CFC/WLC. | Pre to post individual CBT (estimated up to 2 years, depending upon the patient's specific needs)
  Course of depressive symptoms during individual CBT after ART/CFC/WLC. Testing the hypothesis that fostering emotion regulation skills may enhance the efficacy of subsequent individual cognitive behavioral therapy for depression

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Berking, Prof. Dr., Principal Investigator — Friedrich-Alexander-University Erlangen-Nuremberg
Locations (3):
- Germany (3):
  - Philipps-University of Marburg, Marburg, Hesse
  - Aus- und Weiterbildungszentrum für Klinische Verhaltenstherapie, Kassel
  - University of Mainz, Mainz

IPD SHARING:
Plan to Share IPD: Yes
Deidentified IPD will be made available to other researchers upon reguest.
Supporting Information: ICF, Analytic Code
Time Frame: From January 2018 to January 2028
Access Criteria: Credible and legitimate reason for request

REFERENCES:
- [Derived] Eichler E, Hager M, Baeuml J, Berking M. Emotion regulation as mechanism of change in the treatment of depression - A latent change score analysis. J Affect Disord. 2026 Jan 1;392:120205. doi: 10.1016/j.jad.2025.120205. Epub 2025 Sep 2. PMID 40907712
- [Derived] Berking M, Eichler E, Luhmann M, Diedrich A, Hiller W, Rief W. Affect regulation training reduces symptom severity in depression - A randomized controlled trial. PLoS One. 2019 Aug 29;14(8):e0220436. doi: 10.1371/journal.pone.0220436. eCollection 2019. PMID 31465443
- [Derived] Ehret AM, Kowalsky J, Rief W, Hiller W, Berking M. Reducing symptoms of major depressive disorder through a systematic training of general emotion regulation skills: protocol of a randomized controlled trial. BMC Psychiatry. 2014 Jan 27;14:20. doi: 10.1186/1471-244X-14-20. PMID 24467807
- Available data/document: Individual Participant Data Set — https://osf.io/426pd
- Available data/document: All study files — https://osf.io/uhwnb